CLINICAL TRIAL: NCT07154797
Title: A Prospective Trial to Evaluate the Safety and Effectiveness of the Sustained Release Bimatoprost Implant With SpyGlass IOL in Patients With Ocular Hypertension or Mild to Moderate Open-Angle Glaucoma
Brief Title: Evaluation of the Safety and Effectiveness of the Bimatoprost Implant System / IOL Combination in Patients With Ocular Hypertension or Mild to Moderate Open-angle Glaucoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SpyGlass Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SGP-SPEC-001
Record Dates: First submitted 2025-08-22; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Cataract; Ocular Hypertension; Glaucoma
MeSH Terms: conditions — Cataract; Ocular Hypertension; Glaucoma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Bimatoprost Implant System / IOL Combination Low Dose (Experimental): Bimatoprost Implant System (Low Dose) used in combination with the SpyGlass Intraocular Lens
  Interventions: Combination Product: Bimatoprost Implant System / IOL Combination
- Bimatoprost Implant System / IOL Combination Medium Dose (Experimental): Bimatoprost Implant System (Medium Dose) used in combination with the SpyGlass Intraocular Lens
  Interventions: Combination Product: Bimatoprost Implant System / IOL Combination
- Bimatoprost Implant System / IOL Combination High Dose (Experimental): Bimatoprost Implant System (High Dose) used in combination with the SpyGlass Intraocular Lens
  Interventions: Combination Product: Bimatoprost Implant System / IOL Combination

INTERVENTIONS:
Combination Product: Bimatoprost Implant System / IOL Combination — Bimatoprost Implant System used in combination with the SpyGlass intraocular lens

SUMMARY:
The goal of this clinical trial is to learn if the SpyGlass Pharma Bimatoprost Implant System / IOL Combination works to treat cataracts and either ocular hypertension or glaucoma. It will also learn about the safety of the Bimatoprost Implant System / IOL Combination. The main questions it aims to answer are:

* Does the Bimatoprost Implant System / IOL Combination lower the pressure inside the eye to treat ocular hypertension or glaucoma?
* Does the Bimatoprost Implant System / IOL Combination correct vision after cataract surgery?
* What medical problems do participants have when treated with the Bimatoprost Implant System / IOL Combination?

Participants will:

* Upon providing informed consent and successfully completing the screening visit, stop taking their IOP lowering medications in the eye to be treated.
* Complete a baseline visit to further evaluate eligibility in the study eye.
* Undergo standard of care cataract surgery followed by implantation of the Bimatoprost Implant System / IOL Combination. Only one eye of each participant will be treated.
* Complete post-operative follow-up visits for evaluation at Day 1, Week 1, Month 1, Month 3, and Month 6 (last study visit).

DETAILED DESCRIPTION:
This is a single center, proof-of-concept, nonrandomized, multi-arm, controlled clinical trial with a 6-month participation period. The study consists of 3 cohorts of up to 10 participants each. Participants are assigned sequentially to cohorts using a nonrandomized intervention model. Participants will receive standard-of-care cataract extraction by phacoemulsification followed by implantation of the SpyGlass Bimatoprost Implant System / IOL Combination (low-dose cohort; medium-dose cohort; and high-dose cohort). The primary endpoint was measured at 6 months. There was no masking in the study design, however, a 2-person reading method was used for all IOP measurements, wherein Observer 1 adjusts the dial and is masked to the reading on the dial and Observer 2 reads and records the value on the source documentation. Participants in this clinical study are seen for the following visits: a Screening visit, an Eligibility visit (Baseline), a Day 0 or Surgery visit, and postoperative visits at Day 1, Week 1, Month 1, Month 3, and Month 6 (Figure 1). Each participant has one eye designated as the study eye.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of mild to moderate open-angle glaucoma or ocular hypertension
* Planned removal of cataract
* Diagnosis of mild to moderate open-angle glaucoma or ocular hypertension

Exclusion Criteria:

* Pregnant women as confirmed via urine pregnancy test for women of child-bearing age at screening
* History of incisional/refractive corneal surgery
* Pseudoexfoliation, pigmentary glaucoma, traumatic, uveitic, neovascular, or angle-closure glaucoma, or glaucoma associated with vascular disorders
* Other ocular diseases, pathology, or conditions

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-04-21 (Actual); Primary Completion 2022-12-13 (Actual); Study Completion 2022-12-13 (Actual)

PRIMARY OUTCOMES:
Unmedicated eyes with IOP reduction of ≥20% from Baseline to the Month 6 | From Baseline until the end of post-operative follow-up at Month 6
  The proportion of unmedicated eyes with IOP reduction of ≥ 20% from Baseline to the Month 6 exam.

SECONDARY OUTCOMES:
Mean change in unmedicated IOP from Baseline to Month 6 | From Baseline until the end of post-operative follow-up at Month 6
  Mean change in unmedicated IOP (mmHg) from Baseline to Month 6
Number of topical glaucoma medications | From Screening until the end of post-operative follow-up at Month 6
  Number of topical glaucoma medications used at Screening compared to Month 6

OTHER OUTCOMES:
Adverse Events | From Screening to the end of post-operative follow-up at Month 6
  All adverse events occurring during the conduct of this study will be captured and reported.
Supplementary Safety Parameter - BCDVA | From Screening to the end of post-operative follow-up at Month 6
  Best Corrected Distance Visual Acuity (snellen)
Supplementary Safety Parameter - Slit Lamp Examination | From Screening to the end of post-operative follow-up at Month 6
  Slit Lamp Examination Findings
Supplementary Safety Parameter - Fundus Examination | From Screening until the end of post-operative follow-up at Month 6
  Dilated Fundus Examination Findings
Supplementary Safety Parameter - Pachymetry | From Screening until the end of post-operative follow-up at Month 6
  Mean central corneal thickness (micrometers)
Supplementary Safety Parameter - Specular Microscopy | From Baseline until the end of post-operative follow-up at Month 6
  Endothelial cell density (cells per square millimeter)

CONTACTS AND LOCATIONS:
Overall Officials: Sr. Director, Clinical Affairs, Study Chair — SpyGlass Pharma, Inc.
Locations (1):
- Centro Oftalmológico Robles, Santa Rosa de Copán, Honduras

IPD SHARING:
Plan to Share IPD: No
This is a proof of concept trial (first in human).

REFERENCES:
- [Derived] Tan NE, Katz G, Robles M, Gupta PK, Kahook MY, Sussman G, Yoo P, Radcliffe NM. Prospective Pilot Study of Sustained Release Bimatoprost Implant with SpyGlass Intraocular Lens: 3-Year Results. Ophthalmol Ther. 2026 Feb 1. doi: 10.1007/s40123-026-01313-4. Online ahead of print. PMID 41621045